CLINICAL TRIAL: NCT04619186
Title: Comparison of Diffusion-Weighted MRI and Mammography Alone or Combined Mammography and Ultrasonography for Screening Women With a Personal History of Breast Cancer (DIMRISC-2 Study)
Brief Title: Diffusion-Weighted MRI for Breast Cancer Screening in Women With a Personal History of Breast Cancer
Status: Suspended | Type: Observational
Why Stopped: Protocol setting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: Breast Cancer Screening
Record Dates: First submitted 2020-10-30; First posted 2020-11-06 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women with personal history of breast cancer (PHBC) are at risk of developing second breast cancers in the conserved and contralateral breast. Because early detection of second breast cancers at the asymptomatic phase can improve relative survival by 17-28%, guidelines recommend annual mammography screening in women with PHBC. However, lower sensitivity and higher interval cancer rates are observed in women with a PHBC compared with women without, especially in women 50 years or younger and those with dense breasts. In a multicenter comparison study of 754 women, MRI screening detected 3.8 additional cancers and ultrasonography detected 2.4 additional cancers, and increased sensitivity over mammography alone. However, the use of breast MRI is limited not only by high costs and long examination time but also by high false-positive findings. In addition, the use of intravenous gadolinium-based contrast agent is contraindicated in women with renal impairment or contrast material allergy contrast. Supplemental ultrasonography in patients with PHBC reports lower sensitivity with high interval cancer rate. Thus, there is a need to develop a more safe, accurate, and cost-effective supplemental imaging modality for screening in women with PHBC. Diffusion-weighted (DW) MRI is an unenhanced fast, functional modality that measures the movement of water molecules to create tissue contrast. Breast malignancies exhibit hindered diffusion and appear hyperintense on DW MRI with low apparent diffusion coefficient (ADC) compared to normal surrounding tissue. Multiple studies have shown that the use of DW MRI can significantly reduce the false positives and unnecessary benign biopsy of breast MRI. Several studies have shown that DW MRI has a potential to detect mammography occult breast cancers with less false positives compared to ultrasonography. These observations have led to the consideration of utilizing DW MRI to screen women with PHBC. In Diffusion-weighted MRI for Breast Cancer Screening (DIMRISC-2) study, we hypothesized that the screening performance of high-resolution DW MRI at 3.0 T should be superior to mammography alone or combined mammography and ultrasonography in women with PHBC. In our institution, alternating conventional imaging and DW MRI screening is offered for patients who have undergone breast surgery and at increased risk of an interval second breast cancer.

DETAILED DESCRIPTION:
* Primary objective: to compare the screening performance of DW MRI versus mammography alone or combined mammography and ultrasonography in women with PHBC.
* Secondary objective: to compare the tumor and patient characteristics detected by DW MRI and combined mammography and ultrasonography in women with PHBC.
* This is a prospective, single center, observational cohort study.
* A total of 1694 women will be enrolled in this study.
* Two latest 3.0 T MRI scanners with dedicated 16- or 18-channel bilateral breast coil are used for DW MRI. For DW MRI screening, the high-resolution echo-planar imaging sequence is designed to have an in-plane resolution of 1.3 x 1.3 mm and a slice thickness of 3 mm. Three b values of 0, 800, and 1200 sec/mm2 are used and ADC maps are generated based on the b=0 and 800 sec/mm2 DW MRI data. The DW MRI images are reconstructed into single summation images with maximum-intensity projections (MIPs) in the sagittal and axial planes. In addition, T1-weighted imaging sequence is also obtained with in-plane resolution of 1.0 x 1.0 mm and a slice thickness of 1 mm.
* All patients with PHBC undergo digital two-dimensional mammography and physician-performed whole-breast ultrasonography on the same day. DW MRI and conventional imaging (mammography and ultrasonography) are alternatively scheduled at 6-month intervals and the order has been randomized.
* Mammography alone, combined mammography and ultrasonography, and DW MRI will be interpreted independently according to the Breast Imaging Reporting and Data System (BI-RADS) and likelihood of malignancy (Score range, 0%-100%) by trained radiologists. DW MRI interpretation guidelines to be used in this study are based on both qualitative and quantitative assessments. Radiologists are required to successfully complete a training case series of 100 DW MR studies prior to interpreting the DW MRI.
* A negative examination result is defined as a final assessment BI-RADS category of 1, 2, 3 and a positive examination result is defined as a final assessment BI-RADS category of 4 or 5.
* Biopsies of DW MRI-detected lesions are performed under ultrasonography guidance whenever possible or with MR guidance if there is no correlative ultrasonography finding. Pathology of core or surgical biopsy and 1 year follow up is the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 25 years of age at the time of enrollment
2. Women who underwent breast conservation therapy or mastectomy and at increased risk of an interval second breast cancer (Age <50 at first cancer diagnosis; Breast density BI-RADS category 3 and 4; First degree family history; First breast cancer was an interval cancer or symptomatic presentation; First breast cancer was grade 2, 3 or ER and PR negative)

Exclusion Criteria:

1. Women with signs or symptoms of breast cancer
2. Women who had bilateral mastectomy

4. Women who had known metastatic disease 5. Pregnant or lactating women 6. Women with claustrophobia or metallic foreign body

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent breast conservation therapy or mastectomy and at increased risk of an interval second breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1694 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cancer detection rate (CDR) | Baseline to up to 1 year
  Number of detected cancers (invasive cancer and DCIS) /1000 women

SECONDARY OUTCOMES:
Sensitivity | Baseline to up to 1 year
  Number of positive examinations with a tissue diagnosis of cancer within 1 year/All examinations with tissue diagnosis of cancer within the same period
Specificity | Baseline to up to 1 year
  Number of negative examinations without tissue diagnosis of cancer within 1 year/All examinations without tissue diagnosis of cancer within the same period
Recall rate | Baseline to up to 1 year
  Percentage of women screened with recommendation for further imaging prior to next routine examination
Positive predictive value (PPV) | Baseline to up to 1 year
  PPV1: True positive/True positive + False positive
  * PPV2: Number of biopsy confirmed cancers/total number of recommendations for biopsy.
  * PPV3: Number of biopsy confirmed cancers/total number of biopsies performed
Accuracy | Baseline to up to 1 year
  Proportion of true positive results (both true positive and true negative) in the population
  -The area under the (receiver operating characteristic) curve (AUC)
Interval cancer rate | Baseline to up to 1 year
  Breast cancer diagnosed within 1 year of a negative screening result because of clinical symptoms/1000 women
Characteristics of detected cancers | Baseline to up to 1 year
  Tumor size, type, grade, molecular subtype, and lymph node metastasis
Characteristics of women with DW-MRI detected cancer | Baseline to up to 1 year
  Age, menopausal status, breast density, family history

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, MD, PhD, Study Chair — Seoul National University Hosptial
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Ha SM, Chang JM, Lee SH, Kim ES, Kim SY, Kim YS, Cho N, Moon WK. Detection of Contralateral Breast Cancer Using Diffusion-Weighted Magnetic Resonance Imaging in Women with Newly Diagnosed Breast Cancer: Comparison with Combined Mammography and Whole-Breast Ultrasound. Korean J Radiol. 2021 Jun;22(6):867-879. doi: 10.3348/kjr.2020.1183. Epub 2021 Apr 1. PMID 33856137